CLINICAL TRIAL: NCT06376084
Title: Osimertinib With Chemotherapy as First-line Therapy for Patients With Locally Advanced or Metastatic Epidermal Growth Factor Receptor (EGFR) Mutation-positive Non-Small Cell Lung Cancer (NSCLC): A Multicentre, Observational Study (FOREFRONT)
Brief Title: Osimertinib With Chemotherapy as First-line Therapy for EGFR Mutation-positive NSCLC
Acronym: FOREFRONT
Status: Active, not recruiting | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D5161R00055
Record Dates: First submitted 2024-04-17; First posted 2024-04-19 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-12

CONDITIONS: Carcinoma, Non-Small-Cell Lung; Lung Neoplasms; Respiratory Tract Neoplasms; Thoracic Neoplasms; Neoplasms by Site; Neoplasms; Lung Diseases; Respiratory Tract Diseases; Carcinoma, Bronchogenic; Bronchial Neoplasms
Keywords: Osimertinib; Epidermal Growth Factor Receptor; NSCLC; Non-small cell lung cancer; Observational
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms; Respiratory Tract Neoplasms; Thoracic Neoplasms; Neoplasms by Site; Neoplasms; Lung Diseases; Respiratory Tract Diseases; Carcinoma, Bronchogenic; Bronchial Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

SUMMARY:
To estimate parameters related to clinical outcomes in a real-world seeting, including investigator reported PFS and OS .

DETAILED DESCRIPTION:
The objectives of this study are to assess the effectiveness and safety of Osimertinib combined with chemotherapy in a real-world setting in patients with locally advanced or metastatic, EGFR mutation-positive NSCLC.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Histologically or cytologically documented nonsquamous NSCLC. NSCLC of mixed histology is allowed.
* Stage IIIB or IIIC or Stage IV metastatic NSCLC or recurrent NSCLC (based on the American Joint Committee on Cancer Edition 8) not amenable to curative surgery or definitive chemoradiation.
* EGFR sensitive mutation-positive (Ex19del and/or 21 L858R)
* WHO performance status of 0 to 2 at screening with no clinically significant deterioration in the previous 2 weeks.
* Patients who receive Osimertinib plus chemotherapy as first-line treatment based on physician's medical assessment are eligible (For patients who received prior chemotherapy alone/Osimertinib monotherapy/Osimertinib plus chemotherapy as first-line therapy ahead of enrolment, they are diseases progression-free at the time of enrolment and the duration of prior therapy ≤3 months).
* Patients with asymptomatic CNS metastases or patients who have completed definitive therapy, are not on steroids and have a stable neurological status for at least 2 weeks after completion of the definitive therapy and steroids are allowed.
* Prior adjuvant and neo-adjuvant therapies (chemotherapy, radiotherapy, immunotherapy, biologic therapy, investigational agents), or definitive radiation/chemoradiation with or without regimens including immunotherapy, biologic therapies, investigational agents are permitted as long as treatment was completed at least 12 months prior to the development of recurrent disease.

Exclusion Criteria:

* Spinal cord compression and symptomatic brain metastases
* Past medical history of ILD, drug-induced ILD, radiation pneumonitis that required steroid treatment, or any evidence of clinically active ILD
* Any evidence of severe or uncontrolled systemic diseases, including uncontrolled hypertension and active bleeding diatheses, etc
* Any banned substance in label

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with locally advanced or metastatic, EGFR mutation-positive (Ex19del and/or 21 L858R) NSCLC who receive Osimertinib plus chemotherapy as the first-line therapy based on physician's medical assessment will be enrolled. Approximately 700 patients will be enrolled from about 60 sites in China.
Sampling Method: Probability Sample
Enrollment: 532 (Actual)
Dates: Start 2024-07-23 (Actual); Primary Completion 2028-02-28 (Estimated); Study Completion 2028-02-28 (Estimated)

PRIMARY OUTCOMES:
Real-World Progression Free Survival (rwPFS) | Follow up approximately 36 months after last patient in
  rwPFS is defined as the time from the date of first-line initiation until disease progression or death by investigator report as recorded in the CRF

SECONDARY OUTCOMES:
Chemotherapy regimen | Follow up approximately 36 months after last patient in
  Chemotherapy information i.e. dose, number of induction chemotherapy cycles and duration of chemotherapy maintenance, any dose changes and reasons for these changes and date of last administration will also be recorded.
Duration of chemotherapy (induction and maintenance cycles) | Follow up approximately 36 months after last patient in
  Duration of first-line Osimertinib plus chemotherapy, and duration of initial therapy prior to first-line Osimertinib plus chemotherapy (i.e., prior Osimertinib only, prior chemotherapy only).
Response rate | Follow up approximately 36 months after last patient in
  Response rate (RR) is defined as the percentage of patients with the best response of "responding" by investigator report as recorded in CRF. Patients who discontinue treatment without progression, receive a subsequent therapy, and then respond will not be included as responders in the RR calculation.
Duration of response | Follow up approximately 36 months after last patient in
  DoR: is defined as the time from the date of first documented response until the date of documented progression or death in the absence of disease progression. The end of response should coincide with the date of progression or death from any cause used for the PFS endpoint. The time of the initial response will be defined as the latest of the dates contributing toward the first visit response. If a patient does not progress following a response, then his/her duration of response will use the PFS censoring time as the end point for their DoR calculation.
Overall survival (OS) | Follow up approximately 36 months after last patient in
  OS is defined as the time from the first-line initiation until death due to any cause regardless of whether the patient withdraws from therapy or receives another anti-cancer therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Baohui HAN, Principal Investigator — Shanghai Chest Hospital
Locations (1):
- Research Site, Shanghai, China

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. "Yes", indicates that AZ are accepting requests for IPD, but this does not mean all requests will be approved.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA/PhRMA Data-Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. A Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/

REFERENCES:
- [Derived] Zhang B, Ning F, Liu X, Li N, Wang P, Yao W, Han B, Wang Q, Zhong H. First-line therapy of osimertinib with chemotherapy in Chinese patients with EGFR mutation-positive non-small cell lung cancer: protocol for a multicenter, prospective, observational study. Front Oncol. 2025 Sep 5;15:1625714. doi: 10.3389/fonc.2025.1625714. eCollection 2025. PMID 40978050